CLINICAL TRIAL: NCT05369195
Title: Cerebral Protection in Transcatheter Left Atrial Appendage Occlusion in Patients With Atrial Fibrillation
Brief Title: Cerebral Protection in Transcatheter Left Atrial Appendage Occlusion
Acronym: LAAC-SBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Silesian Centre for Heart Diseases (Other)
Collaborators: Leszek Giec Upper-Silesian Medical Centre (Unknown); Medical University of Silesia (Other); Biostat Sp. z o.o. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LAAC-SBI ver. 3
Record Dates: First submitted 2022-03-15; First posted 2022-05-11 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation; Silent Stroke; Cognitive Impairment; Depression
Keywords: cerebral protection; left atrial appendage occlusion; atrial fibrillation; silent brain ischemia; cognitive impairment; depression
MeSH Terms: conditions — Atrial Fibrillation; Cognitive Dysfunction; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In order to blind the radial artery will also be punctured in control group and an aortography will be performed. Researchers participating in the randomization of patients and in the procedure will not be included in the remaining stages of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAAC with neuroprotection (Experimental): Arm in which is used a transcatheter system to protect the cerebral circulation during the left atrial appendage closure procedures.
  Interventions: Procedure: LAAC procedure with the use of transcatheter cerebral protection system
- LAAC without neuroprotection (Placebo Comparator): Arm in which the left atrial appendage closure procedures are performed without transcatheter cerebral protection.
  Interventions: Procedure: LAAC procedure without the use of transcatheter cerebral protection system

INTERVENTIONS:
Procedure: LAAC procedure with the use of transcatheter cerebral protection system — After aortography the cerebral protection system will be delivered to cerebral arteries through radial access before accessing the left atrium.
  Arms: LAAC with neuroprotection
Procedure: LAAC procedure without the use of transcatheter cerebral protection system — Only the aortography through radial access will be done before accessing the left atrium.
  Arms: LAAC without neuroprotection

SUMMARY:
The study aims to assess the effect of the use of neuroprotection in transcutaneous occlusion of the left atrial appendage in patients with atrial fibrillation on the risk of perioperative silent brain ischemia and associated cognitive impairment and depression.

DETAILED DESCRIPTION:
Introduction: Left atrial appendage occlusion (LAAC) procedure is a method of preventing stroke in patients with atrial fibrillation who cannot use anticoagulants. The number of patients undergoing LAAC treatment tends to increase. LAAC procedures effectively reduce the number of strokes, with a significant reduction in the risk of bleeding compared to oral anticoagulants. However, although LAAC treatments alone have a low risk of perioperative stroke, some patients may experience incidents of silent brain ischemia (SBI). The distant effect of SBI may be cognitive deterioration, the onset of dementia syndromes, as well as depression.

Purpose of the study: The study aims to assess the effect of the use of neuroprotection in transcutaneous occlusion of the left atrial appendage (LAAC) in patients with atrial fibrillation on the risk of perioperative SBI and associated cognitive impairment and depression.

Methodology: The planned study is a prospective, multicentre, randomized, and double-blind intervention trial. Neuroprotection introduced from arterial access will be used in the LAAC treatment study group. In the control group, LAAC treatments will be performed without neuroprotection. Two hundred forty patients are planned to be enrolled with indications for stroke prevention due to atrial fibrillation. The analysis will include data obtained from DW MRI images, neurological evaluation results along with NIHSS-scale scores, results of cognitive evaluation tests (MoCA, COWAT, TMT A&B), and test of mood disorders (HADS Scale), as well as results of the EQ-5D-5L quality of life assessment questionnaire. It is planned to observe patients participating in the study for 24 months after LAAC procedure.

ELIGIBILITY:
Inclusion Criteria:

1. 18 Years and older
2. Subject able to provide signed informed consent.
3. Documented permanent, persistent, or paroxysmal atrial fibrillation
4. CHA2DS2VASc risk of stroke ≥2
5. At least one of the following criteria:

   1. Contraindications to the use of anticoagulants,
   2. HSBLED bleeding risk ≥3

Exclusion Criteria:

1. Serious mental diseases, particularly: dementia syndrome of any etiology, schizophrenia,schizoaffective disorders, bipolar disorder
2. History of ischemic stroke
3. Chronic abuse of alcohol or any other psychoactive substances except for nicotine
4. long-term therapy with benzodiazepines
5. The use of antidepressants in 3 months prior inclusion.
6. Previous infections of the central nervous system, including neuroborreliosis
7. Parkinson's disease
8. Huntington's chorea
9. Creutzfeld-Jakob disease
10. Pick's disease
11. Significant atherosclerosis of the cephalic arteries (> 70% LCCA or the brachiocephalic trunk)
12. Strictures, ectasias, dissection or aneurysms at the exit of the LCCA or the brachiocephalic trunk from the aorta and up to 3 cm above
13. Advancement of vascular changes in DW MRI of the head, grade 3 on the Fazekas scale
14. Presence of a thrombus or tumours of a different nature in the left atrium or its ear
15. Presence of a thrombus in the left ventricle
16. Left atrial appendage anatomy preventing the use of occluders to close the left atrium appendage
17. The presence of mechanical heart valve prostheses
18. The state after the operative closure of the defect in the atrial septum
19. Condition after closing the defect in the interatrial septum with the use of occluders
20. Active infective endocarditis
21. Presence of devices and prostheses that prevent the performance of MRI (pacemakers, clips in the CNS)
22. Status after oesophagal surgery
23. Esophageal diverticula
24. Esophageal varices> grade 3
25. Allergic to contrast agents
26. A contraindication to use antiplatelet drugs
27. Diagnosis of neoplastic disease with estimated survival beyond 1 year
28. Clininally evident hypothyroidism and hyperthyroidism
29. Klaustrofobia
30. Pregnancy
31. AIDS
32. Participation in other drug research studies
33. The presence of circumstances or any medical condition the Investigator considers problematic for subject inclusion, or test results that may couse problems to provide reliable, acurate to interpretation results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in number of silent cerebral ischemia (SBI) foci | change in the period up to 24 months
  number of SBI foci in DW MRI of the brain
Change in volume of silent cerebral ischemia (SBI) foci | change in the period up to 24 months
  volume SBI foci in DW MRI of the brain

SECONDARY OUTCOMES:
Deterioration of cognitive functions | prior to procedure, discharge (up to 5 days), 90 days, 12 months, 24 months
  Montreal Cognitive Assessment (MoCA) test (scoring 0-30; cut-off value <26)
Deterioration of cognitive functions | prior to procedure, discharge (up to 5 days), 90 days, 12 months, 24 months
  The Trail Making Test Part A and B for Dementia (TMT A&B) - incorrect values: for part A > 70 sec. and for part B> 273 sec.
Development of dementia | prior to procedure, discharge (up to 5 days), 90 days, 12 months, 24 months
  diagnosis made by a specialist neurologist
Occurrence of depressive disorders | prior to procedure, discharge (up to 5 days), 90 days, 12 months, 24 months
  Hemiltona depression scale - 0 to 50 point, the higher the score, the more severe the mood disorder
Presence of embolic material in the filters of the neuroprotection device | during LAAC procedure

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew F Kalarus, Prof., Principal Investigator — Silesian Centre for Heart Diseases in Zabrze
Locations (6):
- Poland (6):
  - Górnośląskie Centrum Medyczne im. prof. Leszka Gieca Śląskiego Uniwesryeteu Medycznego, Katowice
  - Klinika Chorób Serca i Naczyń, Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow
  - I Klinika Kardiologii Katedry Kardiologii UM im. Karola Marcinkowskiego w Poznaniu, Szpital Kliniczny im. Heliodora Święcickiego UM w Poznaniu, Poznan
  - Klinika Kardiologii i Chorób Wewnętrznych, Wojskowy Instytut Medyczny, Warsaw
  - Klinika Choroby Wieńcowej i Strukturalnych Chorób Serca, Narodowy Instytut Kardiologii Stefana kardynała Wyszyńskiego - Państwowy Instytut Badawczy, Warsaw
  - Silesian Centre for HEart Diseases in Zabrze, Zabrze

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Streb W, Lasek-Bal A, Mitrega K, Kowalczyk J, Podolecki T, Kowalska W, Olma A, Sobczyk A, Kalarus Z. Rationale and design of a randomized clinical trial evaluating the efficacy of mechanical neuroprotection in reducing the risk of silent brain infarcts associated with percutaneous left atrial appendage closure: study protocol for a LAAC-SBI trial. Trials. 2023 Nov 23;24(1):749. doi: 10.1186/s13063-023-07766-3. PMID 37996955